CLINICAL TRIAL: NCT01441362
Title: A Comparison of Two Methods for Intubation With Double-lumen Endobronchial Tube to Reduce Laryngeal Injuries
Brief Title: Double-lumen Tube Intubation Technique to Reduce Laryngeal Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_DLT_180
Record Dates: First submitted 2011-09-25; First posted 2011-09-27 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Laryngeal Injuries
Keywords: during double-lumen; tube intubation

ARMS (2):
- 90 degrees rotation (Active Comparator): Double-lumen tube intubation with 90 degrees rotation
  Interventions: Procedure: 90 degrees rotation
- 180 degrees rotation (Experimental): Double-lumen tube intubation with 180 degrees rotation
  Interventions: Procedure: 180 degrees rotation

INTERVENTIONS:
Procedure: 90 degrees rotation — Double-lumen tube intubation with 90 degrees rotation
  Arms: 90 degrees rotation
Procedure: 180 degrees rotation — Double-lumen tube intubation with 180 degrees rotation
  Arms: 180 degrees rotation

SUMMARY:
The purpose of this study is to devise the method to reduce laryngeal injuries during double-lumen tube intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery that require the placement of left-sided double-lumen tubes

Exclusion Criteria:

* Preoperative hoarseness or sore throat
* History of upper airway diseases
* Anticipated difficult airway
* Operation time longer than 6 hours

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
postoperative hoarseness | up to 3 days

SECONDARY OUTCOMES:
postoperative sore throat | up to 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo JH, Kwon TK, Jeon Y, Hong DM, Kim HJ, Bahk JH. Comparison of techniques for double-lumen endobronchial intubation: 90 degrees or 180 degrees rotation during advancement through the glottis. Br J Anaesth. 2013 Nov;111(5):812-7. doi: 10.1093/bja/aet203. Epub 2013 Jun 20. PMID 23794671